CLINICAL TRIAL: NCT05029882
Title: A Phase 1 First in Human Study Evaluating Safety, Pharmacokinetics and Efficacy of ABBV-400 as Monotherapy and in Combination With Bevacizumab in Adult Subjects With Advanced Solid Tumors
Brief Title: Study to Assess Adverse Events and Change in Disease Activity in Adult Participants With Advanced Solid Tumors Receiving Intravenous (IV) ABBV-400 as Monotherapy and in Combination With IV Bevacizumab
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M21-404; 2023-509335-60-00 (Other: EU CT)
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer; Advanced Solid Tumors; Gastroesophageal Adenocarcinoma; Colorectal Cancer
Keywords: Non-Small Cell Lung Cancer; ABBV-400; Advanced Solid Tumors; Gastroesophageal Adenocarcinoma; Colorectal Cancer; MET Amplification; MET Mutation; Trifluridine/Tipiracil; TAS-102; Bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Part 1 (Monotherapy Dose Escalation) (Experimental): Participants with advanced solid tumors will receive escalating doses of ABBV-400.
  Interventions: Drug: ABBV-400
- Part 2i (wtEGFR Non-Small Cell Lung Cancer [NSCLC]) (Experimental): Participants with non-squamous wtEGFR NSCLC will receive ABBV-400 at the Recommended Phase 2 dose (RP2D).
  Interventions: Drug: ABBV-400
- Part 2ii (mutEGFR NSCLC) (Experimental): Participants with non-Squamous mutEGFR NSCLC will receive ABBV-400 at RP2D.
  Interventions: Drug: ABBV-400
- Part 2iii (Squamous NSCLC) (Experimental): Participants with squamous NSCLC will receive ABBV-400 at RP2D.
  Interventions: Drug: ABBV-400
- Part 3 (Gastroesophageal Adenocarcinoma/Gastroesophagel Junct (Experimental): Participants with gastroesophageal adenocarcinoma will receive ABBV-400 at the RP2D.
  Interventions: Drug: ABBV-400
- Part 4 (Colorectal Cancer) (Experimental): Participants with Colorectal Cancer (CRC) will receive ABBV-400 at the RP2D and various dose levels for dose optimization.
  Interventions: Drug: ABBV-400
- Part 5 (MET Amplification) (Experimental): Participants with mesenchymal-epithelial transition proto-oncogene (MET) amplification will receive ABBV-400 at the RP2D and various dose levels for dose optimization.
  Interventions: Drug: ABBV-400
- Part 6 (MET Mutation) (Experimental): Participants with MET mutation will receive ABBV-400 at the RP2D and various dose levels for dose optimization.
  Interventions: Drug: ABBV-400
- Part 7a (Combination Dose Escalation) (Experimental): Participants with CRC will receive escalating doses of ABBV-400 in combination with bevacizumab.
  Interventions: Drug: ABBV-400; Drug: Bevacizumab
- Part 7bi (Combination Dose Optimization Low Dose) (Experimental): Participants with CRC will receive the low dose determined in the dose escalation arm (Part 7a) of ABBV-400 in combination with bevacizumab.
  Interventions: Drug: ABBV-400; Drug: Bevacizumab
- Part 7bii (Combination Dose Optimization High Dose) (Experimental): Participants with CRC will receive the high dose determined in the dose escalation arm (Part 7a) of ABBV-400 in combination with bevacizumab.
  Interventions: Drug: ABBV-400; Drug: Bevacizumab
- Part 7biii (Combination Comparator) (Experimental): Participants with CRC will receive trifluridine/tipiracil (TAS-102) in combination with bevacizumab.
  Interventions: Drug: Trifluridine/Tipiracil; Drug: Bevacizumab

INTERVENTIONS:
Drug: ABBV-400 — Intravenous (IV) Infusion
  Arms: Part 1 (Monotherapy Dose Escalation); Part 2i (wtEGFR Non-Small Cell Lung Cancer [NSCLC]); Part 2ii (mutEGFR NSCLC); Part 2iii (Squamous NSCLC); Part 3 (Gastroesophageal Adenocarcinoma/Gastroesophagel Junct; Part 4 (Colorectal Cancer); Part 5 (MET Amplification); Part 6 (MET Mutation); Part 7a (Combination Dose Escalation); Part 7bi (Combination Dose Optimization Low Dose); Part 7bii (Combination Dose Optimization High Dose)
Drug: Trifluridine/Tipiracil — Oral Tablet
  Other Names: TAS-102
  Arms: Part 7biii (Combination Comparator)
Drug: Bevacizumab — IV Infusion
  Arms: Part 7a (Combination Dose Escalation); Part 7bi (Combination Dose Optimization Low Dose); Part 7bii (Combination Dose Optimization High Dose); Part 7biii (Combination Comparator)

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess adverse events and change in disease activity when ABBV-400 is given to adult participants to treat advanced solid tumors.

ABBV-400 is an investigational drug being developed for the treatment of advanced solid tumors. Study doctors put the participants in groups called treatment arms. The Recommended Phase 2 dose (RP2D) will be explored. Each treatment arm receives a different dose of ABBV-400. This study will include a dose escalation phase to determine the best dose of ABBV-400, followed by a dose expansion phase to confirm the dose and combination with bevacizumab. Approximately 500 adult participants with NSCLC, gastroesophageal adenocarcinoma/gastroesophagel junction adenocarcinoma (GEA) and colorectal cancer (CRC) or advanced solid tumors, will be enrolled in the study in approximately 7-10 sites in the Dose Escalation phase and 85-95 sites in the Dose Expansion phase worldwide.

Dose escalation arms, participants will receive intravenous (IV) escalating doses of ABBV-400 monotherapy. Dose expansion arms, participants in the following advanced solid tumor indications: non-squamous NSCLC with wildtype EGFR-expression (wtEGFR NSCLC) [Part 2i] or mutated EGFR-expression (mutEGFR NSCLC) [Part 2ii], squamous NSCLC [Part 2iii], GEA [Part 3] will receive intravenous (IV) ABBV-400 monotherapy, participants CRC will receive IV ABBV-400 monotherapy in expansion [Part 4], participants MET amplification will receive IV ABBV-400 monotherapy in expansion [Part 5], participants MET mutation will receive IV ABBV-400 monotherapy in expansion [Part 6], participants CRC safety lead in will receive escalating doses of IV ABBV-400 in combination with IV bevacizumab [Part 7a], and participants CRC dose optimization in will the low or high dose of IV ABBV-400 determined in Part 7a in combination with IV bevacizumab or oral trifluridine/tipiracil (TAS-102) tablets [Part 7b].

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant solid tumor (World Health Organization [WHO] criteria).
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* For Part 1 only - advanced solid tumors including (but not limited to) non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), gastroesophagel junction adenocarcinoma (GEA), colorectal cancer (CRC), and renal cell carcinoma (RCC), who have progressed on all standard of care therapy and are not amenable to surgical resection or other approved therapeutic options that have demonstrated clinical benefit.
* For Part 2 only - advanced non-squamous squamous Non-Small Cell Lung Cancer (NSCLC) that have progressed after treatment with at least:

  * Platinum-based chemotherapy and an immune checkpoint inhibitor and/or appropriate targeted therapy for an actionable gene alteration, if applicable, for non-squamous wtEGFR NSCLC (Part 2i) and squamous NSCLC (Part 2iii).
  * Platinum-based chemotherapy doublet and tyrosine kinase inhibitor(s) (TKI[s]) for non- squamous mutEGFR NSCLC (Part 2ii).
  * Must have no more than 2 lines of prior cytotoxic chemotherapy excluding adjuvant therapy and must have advanced NSCLC that is not amenable to surgical resection or other approved therapeutic options that have demonstrated clinical benefit.
* For Part 3 only - Participants with advanced GEA that has progressed after treatment with at least 1 prior cytotoxic chemotherapeutic regimen for locally advanced or metastatic disease and have not received more than 2 prior lines of cytotoxic chemotherapy regimens. Participants must have progressed on

  * If applicable, an immune checkpoint inhibitor.
  * If applicable, appropriate available therapies, including HER2-directed therapies.

Participants who are considered ineligible for or are intolerant of standard therapy per investigator are eligible.

* For Part 4 only - Participants with history of advanced histopathologically or cytologically confirmed colorectal cancer (CRC) that does not harbor the BRAF V600E mutation and are not dMMR+/MSI-Hi with progression on:

  * A fluoropyrimidine (e.g., 5-fluorouracil or capecitabine).
  * Oxaliplatin.
  * Irinotecan.
  * If applicable, anti-EGFR (including, but not limited to cetuximab or panitumumab).
  * If applicable, anti-vascular endothelial growth factor (VEGF) monoclonal antibody (including but not limited to bevacizumab, ramucirumab, or aflibercept).
  * If applicable, targeted therapy
  * Participants who are considered ineligible for or are intolerant of standard therapy per investigator are eligible. Prior trifluridine/tipiracil (TAS-102) or Regorafenib treated participants are eligible.
* For Part 5 only - participants with advanced histologically or cytologically confirmed solid tumors characterized by MET amplification who are not amenable to surgical resection and who have disease progression after at least one prior systemic therapy and/or who have no satisfactory alternative treatment options. Participants who are intolerant to standard treatment are eligible.

For Part 6 only - Participants with advanced histologically or cytologically confirmed solid tumors harboring MET mutations including: mutations in the tyrosine kinase domain, the juxtamembrane region and the extracellular domain (as locally determined by next-generation sequencing (NGS) or a validated qPCR on tissue), who are not amenable to surgical resection and who have disease progression after at least one prior systemic therapy and/or who have no satisfactory alternative treatment options.

* Intolerant to the standard treatment are eligible
* For Part 7 (CRC combination) only: Participants with history of advanced histopathologically or cytologically confirmed CRC that does not harbor the mutation and are not dMMR+/MSI-H with progression on:

  * A fluoropyrimidine (e.g., 5-fluorouracil or capecitabine)
  * Oxaliplatin
  * Irinotecan
  * If applicable, anti-EGFR (including, but not limited to cetuximab or panitumumab)
  * If applicable, anti-vascular endothelial growth factor (VEGF) monoclonal antibody (including but not limited to bevacizumab, ramucirumab, or aflibercept)
  * If applicable, targeted therapy Participants who are considered ineligible for or are intolerant of standard therapy per investigator are eligible. Participants treated previously with TAS-102 or regorafenib are not eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Laboratory values meeting the criteria outlined in the protocol.

Exclusion Criteria:

* History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, nor any evidence of active ILD or on screening chest CT scan..
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis.
* History of clinically significant, intercurrent lung-specific illnesses, as noted in the protocol.
* For Part 7 only: Prior TAS-102 or regorafenib treated participants are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 48 Months
  ORR defined as percentage of participants with confirmed best overall response of Confirmed complete response (CR) and partial response (PR) per investigator review according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Duration of Response (DOR) for Participants with Confirmed CR/PR per RECIST v1.1 | Up to 48 Months
  DOR is defined for participants achieving a confirmed CR+PR as the time from the initial response of CR+PR per investigator review according to RECIST 1.1 criteria to disease progression or death of any cause, whichever occurs earlier.
PFS per RECIST v1.1 | Up to 48 Months
  Progression-free survival (PFS) is defined as time from first study treatment to a documented disease progression according to RECIST version 1.1, as determined by the investigator, or death due to any cause, whichever occurs earlier.
Overall survival (OS) | Up to 48 Months
  Overall survival (OS) is defined as time from first study treatment to death due to any cause.
Parts 1-6: ORR per Independent Central Review (ICR) in Participants with MET Amplification | Up to 48 Months
  ORR defined as percentage of participants with confirmed best overall response of confirmed CR and PR per ICR according to RECIST version 1.1 in participants with MET amplification.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (82):
- United States (18):
  - University of California, Los Angeles /ID# 243841, Los Angeles, California
  - University Of Colorado Denver /ID# 231574, Aurora, Colorado
  - Yale School of Medicine /ID# 248418, New Haven, Connecticut
  - University of Illinois Hospital and Health Sciences System /ID# 251386, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology - Fort Wayne - East Dupont Road /ID# 267338, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center /ID# 245133, Indianapolis, Indiana
  - Community Health Network, Inc. /ID# 245331, Indianapolis, Indiana
  - Comprehensive Cancer Centers of Nevada /ID# 242930, Henderson, Louisiana
  - START Midwest /ID# 231551, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 250668, New York, New York
  - Duke Cancer Institute /ID# 247236, Durham, North Carolina
  - Carolina BioOncology Institute /ID# 231541, Huntersville, North Carolina
  - Duplicate_Gabrail Cancer Center Research /ID# 248419, Canton, Ohio
  - MD Anderson Cancer Center at Texas Medical Center /ID# 248656, Houston, Texas
  - Oncology Consultants /ID# 267347, Houston, Texas
  - NEXT Oncology /ID# 231578, San Antonio, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 231575, Fairfax, Virginia
  - Northwest Medical Specialties Tacoma /ID# 267339, Tacoma, Washington
- Australia (2):
  - Mater Misericordiae Limited /ID# 249995, South Brisbane, Queensland
  - Austin Health /ID# 247667, Heidelberg, Victoria
- France (8):
  - Institut Bergonie /ID# 248028, Bordeaux, Gironde
  - CHU Nantes - Hopital Laennec /ID# 244723, Saint-Herblain, Loire-Atlantique
  - Institut de Cancérologie de l'Ouest René Gauducheau /ID# 248399, Saint-Herblain, Loire-Atlantique
  - Centre Antoine-Lacassagne /ID# 231730, Nice, Provence-Alpes-Côte d'Azur Region
  - Centre Leon Berard /ID# 250987, Lyon, Rhone
  - Institut Gustave Roussy /ID# 246824, Villejuif, Val-de-Marne
  - Centre Georges François Leclerc /ID# 244450, Dijon
  - AP-HP - Hopital Européen Georges Pompidou /ID# 250481, Paris
- Israel (6):
  - Meir Medical Center /ID# 244179, Kfar Saba, Central District
  - Hadassah Medical Center /ID# 243821, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 231217, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 245271, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 231218, Haifa
  - Rabin Medical Center /ID# 243363, Petah Tikva
- Japan (10):
  - NHO Nagoya Medical Center /ID# 250286, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 250284, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 232008, Kashiwa-shi, Chiba
  - Yokohama Municipal Citizen's Hospital /ID# 248842, Yokohama, Kanagawa
  - Kyoto University Hospital /ID# 250291, Kyoto, Kyoto
  - Niigata University Medical & Dental Hospital /ID# 250952, Niigata, Niigata
  - National Cancer Center Hospital /ID# 232007, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 248447, Koto-ku, Tokyo
  - Wakayama Medical University Hospital /ID# 250283, Wakayama, Wakayama
  - Nagasaki University Hospital /ID# 250290, Nagasaki
- Poland (4):
  - Med Polonia Sp. z o. o. /ID# 250799, Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Bada /ID# 246569, Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio /ID# 251846, Przemyśl, Podkarpackie Voivodeship
  - Samodzielny Publiczny Zespó? Gru?licy i Chorób P?uc w Olsztynie /ID# 250466, Olsztyn
- Pan American Center for Oncology Trials, LLC /ID# 231580, Rio Piedras, Puerto Rico
- South Korea (10):
  - Inje University Haeundae Hospital /ID# 244451, Busan, Busan Gwang Yeogsi
  - CHA Bundang Medical Center /ID# 247115, Seongnam, Gyeonggido
  - Gyeongsang National University Hospital /ID# 248420, Jinju, Gyeongsangnam-do
  - Chungbuk National University Hospital /ID# 245168, Cheongju-si, North Chungcheong
  - Seoul National University Hospital /ID# 244667, Seoul, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 248401, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 245215, Seoul, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 248421, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital /ID# 244504, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 245218, Seoul
- Spain (13):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 245378, Santiago de Compostela, A Coruna
  - Instituto Catalan de Oncologia (ICO) Badalona /ID# 245379, Badalona, Barcelona
  - Hospital Universitario Fundacion Alcorcon /ID# 244505, Alcorcón, Madrid
  - Clinica Universidad de Navarra - Pamplona /ID# 248816, Pamplona, Navarre
  - Hospital Universitario Vall de Hebron /ID# 249809, Barcelona
  - Hospital Clinic de Barcelona /ID# 245374, Barcelona
  - Hospital Universitario de Jaen /ID# 249201, Jaén
  - Hospital General Universitario Gregorio Maranon /ID# 245270, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 231464, Madrid
  - Hospital Universitario 12 de Octubre /ID# 248417, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 244721, Madrid
  - Hospital Universitario Virgen Macarena /ID# 245213, Seville
  - Hospital Universitario Miguel Servet /ID# 244456, Zaragoza
- Taiwan (10):
  - Duplicate_Kaohsiung Chang Gung Memorial Hospital /ID# 246449, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 245731, Taipei City, Taipei
  - Changhua Christian Hospital /ID# 249150, Changhua City, Changhua County
  - Cmuh /Id# 245729, Taichung
  - National Cheng Kung University Hospital /ID# 245918, Tainan
  - Taipei Medical University Hospital /ID# 245732, Taipei
  - Taipei Veterans General Hosp /ID# 250652, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center /ID# 245917, Taipei
  - Tri-Service General Hospital /ID# 245733, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 248716, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-404